CLINICAL TRIAL: NCT01583686
Title: Phase I/II Study of Metastatic Cancer Using Lymphodepleting Conditioning Followed by Infusion of Anti-mesothelin Gene Engineered Lymphocytes
Brief Title: CAR T Cell Receptor Immunotherapy Targeting Mesothelin for Patients With Metastatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to slow/insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 120111; 12-C-0111
Record Dates: First submitted 2012-04-20; First posted 2012-04-24 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Cervical Cancer; Pancreatic Cancer; Ovarian Cancer; Mesothelioma; Lung Cancer
Keywords: Metastatic Cancer; Immunotherapy; Gene Therapy; Mesothelioma; Pancreatic Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Mesothelioma; Lung Neoplasms; Neoplasm Metastasis | interventions — fludarabine; fludarabine phosphate; Automobiles; Cyclophosphamide; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I (Experimental): Non-myeloablative but lymphodepleting preparative regimen of cyclophosphamide and fludarabine plus anti-mesothelin chimeric T cell receptor (CAR) transduced peripheral blood lymphocytes (PBL) plus low dose aldesleukin.
  Interventions: Drug: Fludarabine; Biological: Anti-mesothelin chimeric T cell receptor (CAR) transduced peripheral blood lymphocytes (PBL); Drug: Cyclophosphamide; Drug: Aldesleukin
- 2/Phase II (Experimental): Non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine + anti-mesothelin chimeric T cell receptor (CAR) transduced peripheral blood lymphocytes (PBL) + low-dose aldesleukin
  Interventions: Drug: Fludarabine; Biological: Anti-mesothelin chimeric T cell receptor (CAR) transduced peripheral blood lymphocytes (PBL); Drug: Cyclophosphamide; Drug: Aldesleukin

INTERVENTIONS:
Drug: Fludarabine — Days -5 to Day -1: Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Biological: Anti-mesothelin chimeric T cell receptor (CAR) transduced peripheral blood lymphocytes (PBL) — Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20 to 30 minutes.
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml 5% dextrose in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Other Names: Cytoxan
Drug: Aldesleukin — Aldesleukin 72,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
  Other Names: Proleukin

SUMMARY:
Background:

The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy for treating patients with metastatic cancer that involves taking white blood cells from the patient, growing them in the laboratory in large numbers, genetically modifying these specific cells with a type of virus (retrovirus) to attack only the tumor cells, and then giving the cells back to the patient. This type of therapy is called gene transfer. In this protocol, we are modifying the patients white blood cells with a retrovirus that has the gene for anti-mesothelin incorporated in the retrovirus.

Objective:

The purpose of this study is to determine a safe number of these cells to infuse and to see if these tumor fighting cells (anti-mesothelin cells) cause metastatic cancer tumors to shrink.

Eligibility:

- Adults age 18-70 with metastatic cancer expressing the mesothelin molecule.

Design:

Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed

Leukapheresis: If the patients meet all of the requirements for the study they will undergo leukapheresis to obtain white blood cells to make the anti-mesothelin cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}

Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the anti-mesothelin cells, and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.

Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits will take up to 2 days.

DETAILED DESCRIPTION:
Background:

* We have constructed a single retroviral vector that contains a chimeric T cell receptor (CAR) that recognizes mesothelin, which can be used to mediate genetic transfer of this CAR with high efficiency (> 50%) without the need to perform any selection.
* In co-cultures with mesothelin expressing cells, anti-mesothelin transduced T cells secreted significant amounts of interferon (IFN)-gamma with high specificity.

Objectives:

Primary Objectives:

* To evaluate the safety of the administration of anti-mesothelin CAR engineered peripheral blood lymphocytes in patients receiving a non- myeloablative conditioning regimen, and aldesleukin.
* Determine if the administration anti-mesothelin CAR engineered peripheral blood lymphocytes and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic cancer.

Eligibility:

Patients who are 18 years of age or older must have

* Metastatic or unresectable cancer that expresses mesothelin;
* Previously received and have been a non-responder to or recurred after standard care;

Patients may not have:

-Contraindications for low dose aldesleukin administration.

Design:

* Peripheral blood mononuclear cells (PBMC) obtained by leukapheresis will be cultured in order to stimulate T-cell growth.
* Transduction is initiated by exposure of approximately 10^8 to 5 X 10^8 cells to retroviral vector supernatant containing the anti-mesothelin CAR.
* Patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo CAR gene-transduced PBMC plus low dose intravenous (IV) aldesleukin
* Patients will undergo complete evaluation of tumor with physical examination, Computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment. If the patient has stable disease (SD) or tumor shrinkage, repeat complete evaluations will be performed every 1-3 months. After the first year, patients continuing to respond will continue to be followed with this evaluation every 3-4 months until off study criteria are met.
* The study will be conducted using a Phase I/II optimal design. The protocol will proceed in a phase 1 dose escalation design. Once the maximum tolerated dose (MTD) has been determined, the study then would proceed to the phase II portion. Patients will be entered into two cohorts based on histology: cohort 1 will include patients with mesothelioma, and cohort 2 will include patients with other types of cancer that express mesothelin.
* For each of the 2 strata evaluated, the study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. For each of these two arms of the trial, if 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled in that stratum.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic or unresectable measurable cancers that express mesothelin. As in other protocols conducted by Dr. Hassan in the National Cancer Institute (NCI), epithelial mesotheliomas and pancreatic cancers do not need to be assessed for mesothelin expression since all of these tumors have been shown to express mesothelin. Other metastatic or unresectable cancers must be shown to expresses mesothelin as assessed by reverse transcription polymerase chain reaction (RT-PCR) or immunohistochemistry on tumor tissue. Bi-phasic mesotheliomas must express mesothelin on greater than 50% of the cells in the epithelial component. Diagnosis will be confirmed by the Laboratory of Pathology, NCI.
  2. Patients must have previously received at least one systemic standard care (or effective salvage chemotherapy regimens) for metastatic or unresectable disease, if known to be effective for that disease, and have been either non-responders (progressive disease) or have recurred.
  3. Greater than or equal to 18 years of age and less than or equal to 70 years of age.
  4. Willing to sign a durable power of attorney
  5. Able to understand and sign the Informed Consent Document
  6. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  7. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
  8. Serology:

     1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
     2. Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be Hepatitis C virus ribonucleic acid (HCV RNA) negative.
  9. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
  10. Hematology:

      1. Absolute neutrophil count greater than 1000/mm(3) without the support of filgrastim.
      2. White blood cell (WBC) (> 3000/mm(3)).
      3. Platelet count greater than 100,000/mm(3).
      4. Hemoglobin greater than 8.0 g/dl.
  11. Chemistry:

      1. Serum alanine aminotransferase/aspartate aminotransferase (ALT/AST) less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  12. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patient's toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

      Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.
  13. Subject's must be co-enrolled in protocol 03-C-0277.

EXCLUSION CRITERIA:

1. Patients with sarcomatoid mesothelioma as mesothelin is not expressed in this type of mesothelioma.
2. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
3. Patients with known brain metastases.
4. Patients receiving full dose anticoagulative therapy.
5. Active systemic infections (e.g.: requiring anti-infective treatment), coagulation disorders or any other major medical illnesses.
6. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
7. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
8. Patients with diabetic retinopathy.
9. Concurrent Systemic steroid therapy.
10. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
11. History of coronary revascularization or ischemic symptoms.
12. Documented left ventricular ejection fraction (LVEF) of less than or equal to 45% tested in patients with:

    * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second- or third-degree heart block, chest pain, or ischemic heart disease
    * Age greater than or equal to 65 years old
13. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

    * A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
    * Symptoms of respiratory dysfunction
14. Patients who are receiving any other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05-04 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan R, Bullock S, Premkumar A, Kreitman RJ, Kindler H, Willingham MC, Pastan I. Phase I study of SS1P, a recombinant anti-mesothelin immunotoxin given as a bolus I.V. infusion to patients with mesothelin-expressing mesothelioma, ovarian, and pancreatic cancers. Clin Cancer Res. 2007 Sep 1;13(17):5144-9. doi: 10.1158/1078-0432.CCR-07-0869. PMID 17785569
- [Background] Chang K, Pai LH, Pass H, Pogrebniak HW, Tsao MS, Pastan I, Willingham MC. Monoclonal antibody K1 reacts with epithelial mesothelioma but not with lung adenocarcinoma. Am J Surg Pathol. 1992 Mar;16(3):259-68. doi: 10.1097/00000478-199203000-00006. PMID 1599018
- [Background] Hassan R, Cohen SJ, Phillips M, Pastan I, Sharon E, Kelly RJ, Schweizer C, Weil S, Laheru D. Phase I clinical trial of the chimeric anti-mesothelin monoclonal antibody MORAb-009 in patients with mesothelin-expressing cancers. Clin Cancer Res. 2010 Dec 15;16(24):6132-8. doi: 10.1158/1078-0432.CCR-10-2275. Epub 2010 Oct 29. PMID 21037025

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All reporting groups are in the Phase I portion of the study because the study was terminated before reaching phase II.
Groups:
- Arm A01 Anti-mesothelin CAR PBL 1x10^6 + IL-2; Arm A02 Anti-mesothelin CAR PBL 3x10^6 + IL-2; Arm A03 Anti-mesothelin CAR PBL 1x10^7 + IL-2; Arm A04 Anti-mesothelin CAR PBL 3x10^7 + IL-2; Arm A05 Anti-mesothelin CAR PBL 1x10^8 + IL-2: 1/Phase I:
  Drug: Fludarabine
  Days -5 to Day -1: Fludarabine 25 mg/m^2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days.
  Other Names: •Fludara
  Biological/Vaccine: Anti-mesothelin chimeric T cell receptor (CAR) transduced peripheral blood lymphocytes (PBL)
  Day 0: Cells will be infused intravenously (IV) on the Patient Care Unit over 20 to 30 minutes.
  Drug: Cyclophosphamide
  Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml 5% dextrose in water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Other Names: •Cytoxan
  Drug: Aldesleukin
  Aldesleukin 72,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
  Other Names: •Proleukin
Period: Overall Study
Arm/Group | Arm A01 Anti-mesothelin CAR PBL 1x10^6 + IL-2 | Arm A02 Anti-mesothelin CAR PBL 3x10^6 + IL-2 | Arm A03 Anti-mesothelin CAR PBL 1x10^7 + IL-2 | Arm A04 Anti-mesothelin CAR PBL 3x10^7 + IL-2 | Arm A05 Anti-mesothelin CAR PBL 1x10^8 + IL-2
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A01 Anti-mesothelin CAR PBL 1x10^6 + IL-2 | Arm A02 Anti-mesothelin CAR PBL 3x10^6 + IL-2 | Arm A03 Anti-mesothelin CAR PBL 1x10^7 + IL-2 | Arm A04 Anti-mesothelin CAR PBL 3x10^7 + IL-2 | Arm A05 Anti-mesothelin CAR PBL 1x10^8 + IL-2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 3 | 15
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (5.57) | 56.03 (1.6) | 58.4 (1.31) | 51.77 (6.38) | 47.97 (16.1) | 54.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 3 | 3 | 11
  Male | 2 | 1 | 1 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 2
  White | 2 | 3 | 2 | 1 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Tumor Regression
Description: Objective tumor regression response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.0. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum LD. Progressive Disease (PD) is at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 3.5 mos.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A01 Anti-mesothelin CAR PBL 1x10^6 + IL-2 | Arm A02 Anti-mesothelin CAR PBL 3x10^6 + IL-2 | Arm A03 Anti-mesothelin CAR PBL 1x10^7 + IL-2 | Arm A04 Anti-mesothelin CAR PBL 3x10^7 + IL-2 | Arm A05 Anti-mesothelin CAR PBL 1x10^8 + IL-2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0
  Stable Disease | 0 | 1 | 0 | 0 | 0
  Progressive Disease | 3 | 2 | 3 | 3 | 3

2. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 6 months and 17 days for Group A01, 16 months and 13 days for Group A02, 13 months and 3 days for Group A03, 10 months and 16 days for Group A04, and 11 months and 26 days for Group A05.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A01 Anti-mesothelin CAR PBL 1x10^6 + IL-2 | Arm A02 Anti-mesothelin CAR PBL 3x10^6 + IL-2 | Arm A03 Anti-mesothelin CAR PBL 1x10^7 + IL-2 | Arm A04 Anti-mesothelin CAR PBL 3x10^7 + IL-2 | Arm A05 Anti-mesothelin CAR PBL 1x10^8 + IL-2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 3 | 3 | 3 | 3 | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 6 months and 17 days for Group A01, 16 months and 13 days for Group A02, 13 months and 3 days for Group A03, 10 months and 16 days for Group A04, and 11 months and 26 days for Group A05.
Arm/Group | Arm A01 Anti-mesothelin CAR PBL 1x10^6 + IL-2 | Arm A02 Anti-mesothelin CAR PBL 3x10^6 + IL-2 | Arm A03 Anti-mesothelin CAR PBL 1x10^7 + IL-2 | Arm A04 Anti-mesothelin CAR PBL 3x10^7 + IL-2 | Arm A05 Anti-mesothelin CAR PBL 1x10^8 + IL-2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 0/3 | 1/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A01 Anti-mesothelin CAR PBL 1x10^6 + IL-2 (N=3) | Arm A02 Anti-mesothelin CAR PBL 3x10^6 + IL-2 (N=3) | Arm A03 Anti-mesothelin CAR PBL 1x10^7 + IL-2 (N=3) | Arm A04 Anti-mesothelin CAR PBL 3x10^7 + IL-2 (N=3) | Arm A05 Anti-mesothelin CAR PBL 1x10^8 + IL-2 (N=3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A01 Anti-mesothelin CAR PBL 1x10^6 + IL-2 (N=3) | Arm A02 Anti-mesothelin CAR PBL 3x10^6 + IL-2 (N=3) | Arm A03 Anti-mesothelin CAR PBL 1x10^7 + IL-2 (N=3) | Arm A04 Anti-mesothelin CAR PBL 3x10^7 + IL-2 (N=3) | Arm A05 Anti-mesothelin CAR PBL 1x10^8 + IL-2 (N=3)
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Infection with unknown ANC: Nerve-peripheral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Albumin (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia: Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 3 (3)
Neutrophils/granulocytes (ANC/AGC) count decreased (Investigations) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 3 (3)
Platelets (Investigations) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Thrombosis/embolism (vascular access related) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PTT (Partial Thromboplastin Time) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRALI (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phosphate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT01583686/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT01583686/ICF_001.pdf